CLINICAL TRIAL: NCT02896075
Title: Social Laughter's Effect on Pain Tolerance
Brief Title: Mirthful Laughter and Muscle Soreness / Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-05-0092
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pain
Keywords: delayed onset muscle soreness; laughter
MeSH Terms: conditions — Pain; Laughter

STUDY DESIGN:
Intervention Model Description: The main study was conducted using a randomized controlled cross-over approach.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Randomized cross-over approach (Experimental): The main study was conducted using a randomized controlled cross-over approach. Participants made three visits each for the two video watching interventions. The interventions were separated by a minimum of
  1week as a washout. Each intervention included one day of inducing muscle soreness in one leg through eccentric muscle contractions; a second day of testing muscle soreness and pain tolerance and watching a 30-min video (either a comedy or documentary); and a third day of testing muscle soreness and pain tolerance again to see if the effects of the video viewing persisted the next day (i.e., 24 h after the video viewing).
  Interventions: Other: 30 Minute Comedy Video; Other: 30 Minute Documentary Video

INTERVENTIONS:
Other: 30 Minute Comedy Video — The intervention is a 30 minute video of a comedy
Other: 30 Minute Documentary Video — The intervention is a 30 minute video of an uninteresting documentary

SUMMARY:
The purpose of this study is first to investigate the effect of a controlled intervention with a comedy video on pain tolerance in a social setting while quantitatively measuring laughter in a young healthy population experiencing delayed onset muscle soreness. The comedy intervention will be compared to a control of watching a documentary. The second aim is to examine to what extent various methods of eliciting pain would cause physiological responses that confound the interpretation of a pain stimulus.

DETAILED DESCRIPTION:
Chronic pain affects 116 million people, that is more than the total affected by cardiovascular disease, cancer, and diabetes combined. Chronic pain has at least as large of a negative impact on quality of life as any other chronic disorder, and in the United States alone, the cost of chronic pain exceeds $635 billion per year. Interventions that effectively manage chronic pain are becoming increasingly important as the elderly population, who often suffer from osteoarthritis and low back pain, rises. Pain sensitivity and tolerance are impacted by a variety of affective factors. The laughter therapy is one of the most discussed and often controversial strategies for the management of pain. There are some preliminary uncontrolled studies reporting that pain tolerance is increased acutely with humor and laughter. Accordingly, the primary aim of the present study is to investigate the effect of a highly controlled intervention with a comedy video on pain tolerance and compare it to a control of watching a documentary video. Quantitatively measuring laughter with a chest stress-strain gauge during the interventions will allow the investigators to look for a possible dose response relationship. The investigators will use the pain and soreness felt from delayed onset muscle soreness (DOMS) in healthy subjects to simulate the condition of individuals suffering from chronic pain. This study will serve as a precursor to eventual studies specifically on individuals with chronic pain. If it can be proven that pain tolerance is increased in a healthy population than it is possible the intervention will have a greater affect in the chronic pain population.

Using healthy subjects with delayed onset muscle soreness allows the investigators to easily recruit and control for other diseases or disorders that may accompany a chronic pain individual.

There have been a number of different techniques used to assess pain tolerance. The modes of stimulating pain used in previous studies of laughter and humor on pain tolerance remain controversial. These studies utilized the cold pressor test and the inflation of a blood pressure cuff to elicit pain. Both of these methods are known to elicit marked cardiovascular responses along with the pain responses. An important part of the pain regulatory process in humans is that there is a functional interaction between the cardiovascular and pain regulatory systems. The brain regions underlying control of the cardiovascular system are known to overlap substantially with those that contribute to anti-nociception. Accordingly, it is difficult to determine how much of the pain tolerance is affected by cardiovascular reflexes. Thus, the secondary aim of the present study is to test how much cardiovascular responses will be elicited by a variety of methods of eliciting pain (pumping up a blood pressure cuff, the cold pressor test, and the application of blunt force on muscles).

The application of blunt force will be used to elicit pain without causing a systemic response involving cardiovascular reflexes which is seen in the cold pressor and inflation of a blood pressure cuff. The investigators believe these vast cardiovascular responses may cause pain tolerance to not be truly measured. It has been inferred that blunt force applied within a few seconds to a local, specific spot on the quadriceps will not stimulate a systemic and cardiovascular response and thus the pain tolerance measurement will be more accurate if independent of cardiovascular responses. Pressure and force application is widely used as an experimental pain stimulus, but it has not been utilized in the context of laughter and pain.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 20 and 40
* Considered healthy

Exclusion Criteria:

* Candidates that are on cardiovascular acting drugs.
* Candidates currently taking anticoagulants.
* Candidates that have chronic pain or other musculoskeletal injuries.
* Candidates with a body fat percentage less than 5%.
* Candidates with bleeding disorders or neurological disorders
* Raynaud's disease
* History of severe frost bite.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hirofumi Tanaka, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Cardiovascular Aging Research Lab at UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lapierre SS, Baker BD, Tanaka H. Effects of mirthful laughter on pain tolerance: A randomized controlled investigation. J Bodyw Mov Ther. 2019 Oct;23(4):733-738. doi: 10.1016/j.jbmt.2019.04.005. Epub 2019 Apr 13. PMID 31733755

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University student body and the city surrounding the university using flyers
Pre-assignment Details: Each intervention included one day of inducing muscle soreness in one leg through eccentric muscle contractions; a second day of testing muscle soreness and pain tolerance and watching a 30-min video (either a comedy or documentary); and a third day of testing muscle soreness and pain tolerance again to see if the effects of the video viewing persisted the next day (i.e., 24 h after the video viewing).
Groups:
- All Study Participants Acting Their Own Controls: Each intervention included one day of inducing muscle soreness in one leg through eccentric muscle contractions; a second day of testing muscle soreness and pain tolerance and watching a 30-min video (either a comedy or documentary); and a third day of testing muscle soreness and pain tolerance again to see if the effects of the video viewing persisted the next day (i.e., 24 h after the video viewing).
Period: Overall Study
Arm/Group | All Study Participants Acting Their Own Controls
Started | 40
Leg Soreness | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: young healthy people with delayed onset muscle soreness in either the right or left leg will go through the 30 Minute Comedy Video and the 30 Minute Documentary Video.
  30 Minute Comedy Video: The intervention is a 30 minute video of a comedy
  30 Minute Documentary Video: The intervention is a 30 minute video of an uninteresting documentary
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Peak Force of Pain Tolerance Measurement
Description: The peak force is measured by using a force transducer and applying it to participants' quadriceps. Using data acquisition software the investigators can find the peak force applied.
Time Frame: This was measured at 24 hours after watching either a comedy or documentary film.
Measure: Mean (Standard Deviation); unit: N
Groups:
- Comedy Video: The intervention is watching a 30 minute video of a comedy
- Documentary Watching: The intervention is watching a 30 minute video of a documentary
Arm/Group | Comedy Video | Documentary Watching
Number analyzed (Participants) | 40 | 40
N | 2 (3) | 21 (5)

2. Secondary Outcome: Heart Rate
Description: The heart rate was using a finger photoplethysmograph.
Time Frame: This was measured at 24 hours after watching either a comedy or documentary video.
Measure: Mean (Standard Error); unit: beats/minutres
Groups:
- Comedy Watching: The intervention is watching a 30 minute video of a comedy
Arm/Group | Comedy Watching | Documentary Watching
Number analyzed (Participants) | 40 | 40
beats/minutres | 67 (12) | 66 (13)

3. Secondary Outcome: Blood Pressure
Description: Blood pressure on the brachial artery measured via oscillometric methods
Time Frame: This was measured at 24 hours after watching a comedy or documentary video.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Comedy Watching | Documentary Watching
Number analyzed (Participants) | 40 | 40
mmHg
  Systolic blood pressure | 116 (10) | 116 (10)
  Diastolic blood pressure | 57 (7) | 57 (7)

ADVERSE EVENTS:
Time Frame: ~9 months
Description: This is a behavioral observational study that participants were asked to watch videos in the laboratory. No adverse event would be expected.
Groups:
- Leg With and Without Delayed Onset Muscle Soreness: young healthy people with delayed onset muscle soreness in either the right or left leg will go through the 30 Minute Comedy Video and the 30 Minute Documentary Video.
  30 Minute Comedy Video: The intervention is a 30 minute video of a comedy
  30 Minute Documentary Video: The intervention is a 30 minute video of an uninteresting documentary
Arm/Group | Leg With and Without Delayed Onset Muscle Soreness
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT02896075/Prot_SAP_000.pdf